CLINICAL TRIAL: NCT00694551
Title: Pilot Immunotherapy Study of Combination PSMA and TARP Peptide With Poly IC-LC Adjuvant in HLA-A2 (+) Patients With Elevated PSA After Initial Definitive Treatment
Brief Title: PSMA and TARP Peptide Vaccine With Poly IC-LC Adjuvant in HLA-A2 (+) Patients With Elevated PSA After Initial Definitive Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15262; 106346 (Other: USF IRB); 20-14555-05-01 (Other Grant/Funding Number: SPORE in prostate cancer - Pro)
Record Dates: First submitted 2008-06-04; First posted 2008-06-10 (Estimated); Results first posted 2014-02-19 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Prostate Cancer
Keywords: vaccine; PSMA; TARP; immunology; PSA
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Protein Subunit Vaccines; poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A. Level 100 mcg Peptide Vaccine (Experimental): Peptide vaccine dose level 100 mcg + Poly IC-LC
  Interventions: Biological: Peptide Vaccine; Drug: Poly IC-LC
- B. Level 300 mcg Peptide Vaccine (Experimental): Peptide vaccine dose level 300 mcg + Poly IC-LC
  Interventions: Biological: Peptide Vaccine; Drug: Poly IC-LC
- C. Level 1 mg Peptide Vaccine (Experimental): Peptide vaccine dose level 1 mg + Poly IC-LC
  Interventions: Biological: Peptide Vaccine; Drug: Poly IC-LC

INTERVENTIONS:
Biological: Peptide Vaccine — Peptide vaccine (PSMA and TARP peptide vaccine with Poly IC-LC adjuvant). Pilot study using three treatment arms of increasing peptide dose levels (100 mcg, 300 mcg, and 1 mg) with a fixed dose of Poly IC-LC as an adjuvant. Patients were randomly assigned to one of the 3 arms upon enrollment.
  Other Names: Hiltonol; poly IC-LC; PSMA peptide vaccine; TARP peptide vaccine
Drug: Poly IC-LC — Administered subcutaneously, one 2 mg/ml vial,(divided into two equal portions for each injection site).
  Other Names: Hiltonol; NSC-301463

SUMMARY:
Pilot Immunotherapy Study of Combination Prostate Specific Membrane Antigen (PSMA) and T-cell receptor γ alternate reading frame protein (TARP) Peptide With Poly IC-LC Adjuvant in Human Leukocyte Antigens (HLA)-A2 (+) Patients With Elevated prostatic specific antigen (PSA) After Initial Definitive Treatment

The purpose of the study is to see if the PSMA/TARP proteins in the vaccine, along with the Hiltonol, can arouse and train the immune system to kill the prostate cancer cells. Prostate cancer is the most common cancer and is the second leading cause of cancer deaths in U.S. males. It is curable when it is confined to the prostate (kept from spreading) using surgery or radiation treatments. In some patients the cancer can come back after these treatments. Treatment options for prostate cancer that comes back include procedures or medications which may have significant risks and side effects. Another plan is being looked at that uses the body's immune system to attack prostate cancer cells. A vaccine has been developed that has proteins found in prostate cancer cells. One of the proteins is called PSMA and the other is called TARP. In addition to these proteins, another substance called Poly IC-LC (Hiltonol) will be added to the vaccine to boost its ability to start the immune system.

DETAILED DESCRIPTION:
Detailed Objectives:

1. Estimate the frequency of immunological efficacy of the vaccine by comparison of the in vitro enzyme-linked immunosorbent spot (ELISpot) test results, for each antigen (PSMA, TARP) from peripheral blood specimens collected during the periods of time defined as "before", "during" and "after" vaccination.
2. Study the safety and toxicity of varying doses of polypeptide vaccines: PSMA27-35-PSMA687-701 (VLAGGFFLLYRHVIYAPSSHNKYA) and TARP13-35 (LQLLKQSSRRLEHTFMFLRNFSL) administered with a fixed dose of Poly IC-LC (2 mg total/treatment) as adjuvant.
3. Describe the impact of the vaccine on the pattern of PSA change in 2 subsets of patients: with castrate testosterone; with non-suppressed testosterone level/not on hormone therapy.
4. Identify if there is a basis for selection of a dose of the PSMA and the TARP polypeptide vaccines for future phase II development of this vaccination strategy, considering the dose range tested.

ELIGIBILITY:
Inclusion Criteria:

* History of histologically confirmed prostate cancer.
* Competence to understand the patient information and provide written informed consent, and willingness and ability to return to H. Lee Moffitt Cancer Center for planned treatments and follow-up.
* Absence of evidence of metastatic disease by current physical exam or by current imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI] pelvis, and bone scan within 60 days of first treatment).
* Patients not on hormone therapy (stratum "N") must meet all of these:

  1. At least 1 year after prostatectomy, definitive prostate radiation, or other definitive-intent local therapy.
  2. No testosterone suppression therapy for at least 6 months.
  3. PSA at least 1 ng/ml, on 2 measurements, at least 2 weeks apart.
  4. Testosterone level >100 ng/ml, at start ("noncastrate").
* Patients on hormone therapy (stratum "Y") must meet all of these:

  1. On treatment with gonadotropin-releasing hormone (GnRH) agonist (or orchiectomy) at least 6 months.
  2. testosterone level <50 ng/ml, at start.
  3. PSA at least 1 ng/ml, on 2 measurements, at least 2 weeks apart.
* Laboratory values obtained 0-14 days prior to start of therapy:

  1. White blood count (WBC) over 3,500/micro L.
  2. Platelet count over 100,000 micro L.
  3. Hemoglobin over 10.0 g/dL.
  4. Serum creatinine up to 2.0 mg/dL.
  5. Alkaline phosphatase up to 2.5 x upper limit of normal (ULN).
  6. Aspartic transaminase (AST) up to 2.5 x ULN.
* Life expectancy at least 6 months.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.

Exclusion Criteria:

* Known standard therapy for the patient's disease that is potentially curative.
* A known immunodeficiency including HIV. Appropriate trials for individuals with HIV may be considered at a later date.
* History of other malignancy besides prostate cancer in the last 5 years, except non-melanoma skin cancer treated with local resection only. (The effect of study treatment on other, potentially dormant malignant diseases is not known).
* Use of oral or inhaled or parenteral corticosteroids or of other immunomodulatory drugs within the 60 days of start. [Use of steroids after start will be considered by the principal investigator (PI) on a case-by-case basis.]
* Use of estrogens (including herbal phytoestrogens) or ketoconazole within 30 days of start, or during the study.
* Failure to fully recover to grade 1 or better from effects of prior chemotherapy regardless of interval since last treatment.
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or investigational agent in last 30 days (one month washout to start of treatment; patients could register but not start until the washout).
* Known hypersensitivity to one or more components of the study medication.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-12-02 (Actual); Primary Completion 2013-02-28 (Actual); Study Completion 2018-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mayer Fishman, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States
- Ponce School of Medicine, Ponce, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Groups:
- A. Level 100 mcg Peptide Vaccine: Peptide vaccine dose level 100 mcg
  Peptide Vaccine: Peptide vaccine (PSMA and TARP peptide vaccine with Poly IC-LC adjuvant). Pilot study using three treatment arms of increasing peptide dose levels (100 mcg, 300 mcg, and 1 mg) with a fixed dose of Poly IC-LC as an adjuvant. Patients were randomly assigned to one of the 3 arms upon enrollment.
- B. Level 300 mcg Peptide Vaccine: Peptide vaccine dose level 300 mcg
  Peptide Vaccine: Peptide vaccine (PSMA and TARP peptide vaccine with Poly IC-LC adjuvant). Pilot study using three treatment arms of increasing peptide dose levels (100 mcg, 300 mcg, and 1 mg) with a fixed dose of Poly IC-LC as an adjuvant. Patients were randomly assigned to one of the 3 arms upon enrollment.
- C. Level 1 mg Peptide Vaccine: Peptide vaccine dose level 1 mg
  Peptide Vaccine: Peptide vaccine (PSMA and TARP peptide vaccine with Poly IC-LC adjuvant). Pilot study using three treatment arms of increasing peptide dose levels (100 mcg, 300 mcg, and 1 mg) with a fixed dose of Poly IC-LC as an adjuvant. Patients were randomly assigned to one of the 3 arms upon enrollment.
Period: Overall Study
Arm/Group | A. Level 100 mcg Peptide Vaccine | B. Level 300 mcg Peptide Vaccine | C. Level 1 mg Peptide Vaccine
Started | 10 | 10 | 9
Completed | 9 | 10 | 8
Not Completed | 1 | 0 | 1
Not completed — Disease Progression | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All patients who received any amount of study treatment were considered evaluable for toxicity.
Groups:
- A. Peptide Vaccine: Peptide vaccine dose Level 100 mcg
  Peptide Vaccine: Peptide vaccine (PSMA and TARP peptide vaccine with Poly IC-LC adjuvant). Pilot study using three treatment arms of increasing peptide dose levels (100 mcg, 300 mcg, and 1 mg) with a fixed dose of Poly IC-LC as an adjuvant. Patients were randomly assigned to one of the 3 arms upon enrollment.
- B. Peptide Vaccine: Peptide vaccine dose level 300 mcg
  Peptide Vaccine: Peptide vaccine (PSMA and TARP peptide vaccine with Poly IC-LC adjuvant). Pilot study using three treatment arms of increasing peptide dose levels (100 mcg, 300 mcg, and 1 mg) with a fixed dose of Poly IC-LC as an adjuvant. Patients were randomly assigned to one of the 3 arms upon enrollment.
- C. Peptide Vaccine: Peptide vaccine dose level 1 mg
  Peptide Vaccine: Peptide vaccine (PSMA and TARP peptide vaccine with Poly IC-LC adjuvant). Pilot study using three treatment arms of increasing peptide dose levels (100 mcg, 300 mcg, and 1 mg) with a fixed dose of Poly IC-LC as an adjuvant. Patients were randomly assigned to one of the 3 arms upon enrollment.
- Total: Total of all reporting groups
Arm/Group | A. Peptide Vaccine | B. Peptide Vaccine | C. Peptide Vaccine | Total
Number analyzed (Participants) | 10 | 10 | 9 | 29
Age, Continuous [Median (Full Range); unit: years] | 69 [56 to 82] | 69.5 [56 to 83] | 69 [58 to 80] | 69.5 [56 to 83]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 6 | 2 | 9
  >=65 years | 9 | 4 | 7 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 9 | 29
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 9 | 29

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Related Adverse Events - Grade 3 or Higher
Description: Number of participants with related Grade 3 or higher adverse events. Establish the safety and toxicity of varying doses of polypeptide vaccines PSMA and TARP administered with a fixed dose of Poly IC-LC as an adjuvant.
Time Frame: Up to 48 months
Population: All participants who received treatment.
Measure: Number; unit: participants
Arm/Group | A. Level 100 mcg Peptide Vaccine | B. Level 300 mcg Peptide Vaccine | C. Level 1 mg Peptide Vaccine
Number analyzed (Participants) | 10 | 10 | 9
participants | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Prostatic Specific Antigen (PSA) Doubling
Description: Number of Participants Who Had a Doubling of the PSA or Proceeded to Another Therapy.
  Assess the impact of the vaccine on the pattern of PSA change in patients with castrate testosterone level and in patients with non-suppressed testosterone level not on hormone therapy.
Time Frame: Up to 48 months
Population: 29 patients who had serial PSA data, normalized by date and PSA.
Measure: Number; unit: participants
Arm/Group | A. Level 100 mcg Peptide Vaccine | B. Level 300 mcg Peptide Vaccine | C. Level 1 mg Peptide Vaccine
Number analyzed (Participants) | 10 | 10 | 9
participants | 8 | 6 | 5

3. Secondary Outcome: Number of Participants Who Did Not Have PSA Doubling
Description: Number of participants who did not have a PSA doubling before their last study visit, median 458 days from baseline PSA (55-613).
Time Frame: Up to 48 months
Population: 29 patients who had serial PSA data, normalized by date and PSA.
Measure: Number; unit: participants
Arm/Group | A. Level 100 mcg Peptide Vaccine | B. Level 300 mcg Peptide Vaccine | C. Level 1 mg Peptide Vaccine
Number analyzed (Participants) | 10 | 10 | 9
participants | 2 | 4 | 4

ADVERSE EVENTS:
Time Frame: 2 years, 9 months
Arm/Group | A. Peptide Vaccine | B. Peptide Vaccine | C. Peptide Vaccine
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10 | 0/9
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A. Peptide Vaccine (N=10) | B. Peptide Vaccine (N=10) | C. Peptide Vaccine (N=9)
Cough - Grade 2 - (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — PSMA: Unrelated
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A. Peptide Vaccine (N=10) | B. Peptide Vaccine (N=10) | C. Peptide Vaccine (N=9)
Fatigue (General disorders) | 5 (24) | 5 (15) | 6 (29)
Feverr (in the absence of neutropenia) (General disorders) | 6 (17) | 5 (22) | 4 (6)
Rigors/chills (General disorders) | 4 (10) | 6 (18) | 2 (2)
Pain - Head/headache (General disorders) | 3 (15) | 6 (29) | 7 (22)
Pain - Muscle (General disorders) | 4 (11) | 4 (19) | 4 (14)
Pain - Back (General disorders) | 0 (0) | 2 (2) | 3 (3)
Pain - Joint (General disorders) | 3 (3) | 1 (2) | 0 (0)
Pain - Neck (General disorders) | 0 (0) | 2 (2) | 1 (2)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 7 (34) | 9 (46) | 7 (38)
Anorexia (Gastrointestinal disorders) | 2 (3) | 0 (0) | 2 (3)
Nausea (Gastrointestinal disorders) | 2 (4) | 0 (0) | 1 (2)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 4 (9)
Flu-like syndrome (General disorders) | 2 (5) | 1 (1) | 4 (8)
Dizziness (Nervous system disorders) | 2 (4) | 3 (9) | 0 (0)
Lymphatics - Other (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 1 (2)
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 | 0 (0)
Hot flashes/flushes (Endocrine disorders) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes